CLINICAL TRIAL: NCT00063557
Title: Neighborhoods and CVD Risk in a Multiethnic Cohort - Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1220; R01HL071759 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Atherosclerosis

SUMMARY:
To investigate if neighborhood characteristics are related to disease risk in a multiethnic cohort.

DETAILED DESCRIPTION:
BACKGROUND:

Recent epidemiologic studies have found that living in socioeconomically disadvantaged neighborhoods is associated with increased prevalence and incidence of coronary heart disease, even after controlling for measures of personal income, education, and occupation. Although this suggests that features of neighborhoods may be relevant to cardiovascular risk, important questions remain regarding whether the associations observed reflect causal processes. Two important unresolved issues are the role of selection factors in generating these associations and the need to identify the specific characteristics of neighborhoods that are relevant.

DESIGN NARRATIVE:

The study uses publicly available and newly collected neighborhood data linked to the Multi-Ethnic Study of Atherosclerosis (MESA) to: (1) examine the relationship between neighborhood socioeconomic characteristics and the prevalence and progression of subclinical atherosclerosis; (2) examine associations of neighborhood socioeconomic characteristics with specific individual-level factors which may mediate neighborhood differences in disease risk; (3) develop measures of specific characteristics of neighborhood environments (such as measures of resource availability, neighborhood social cohesion and neighborhood stress) and examine their relation to selected individual-level risk factors; (4) determine if these specific neighborhood characteristics explain differences in cardiovascular risk between socioeconomically advantaged and socioeconomically disadvantaged neighborhoods; and (5) examine if neighborhood characteristics contribute to race/ethnic differences in cardiovascular risk. Measures of neighborhood attributes will be based on Year 2000 Census data, surveys of area residents, and the use of GIS methods to link data on area resources to MESA neighborhoods. The examination of subclinical disease as outcomes avoids problems related to selection of persons into neighborhoods based on their health status. The project will use two innovative approaches (residential surveys and ecometric techniques and GIS-based methods) to develop direct measures of specific neighborhood attributes in order to test their relationship to disease risk. Confirming that specific features of neighborhoods are causally related to disease would have important implications for prevention.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Diez-Roux — University of Michigan